CLINICAL TRIAL: NCT03433651
Title: Creatine Monohydrate Use for Preventing Altitude Induced Depression
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to locate grant funding.
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWH20180039H
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depression
Keywords: depression
MeSH Terms: conditions — Depression | interventions — Creatine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Subjects will be randomized using a random number generator to receive either creatine monohydrate or a placebo for 90 days. Both subjects and investigators will be blinded to the study group assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- creatine monohydrate (Experimental): Experimental will take by mouth 5 grams a day of creatine monohydrate powder. Subjects will be given a 30 day supply of the study powder. They will be reminded to take the powder as instructed.
  Interventions: Drug: Creatine monohydrate
- Placebo (Placebo Comparator): Placebo will take by mouth 5 grams a day of placebo powder. Subjects will be given a 30 day supply of the study powder. They will be reminded to take the powder as instructed.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Creatine monohydrate — Subjects will take by mouth 5 grams a day of creatine monohydrate powder.
  Other Names: creapure
  Arms: creatine monohydrate
Drug: Placebo — Subjects will take by mouth 5 grams a day of placebo powder.
  Other Names: maltodextrin
  Arms: Placebo

SUMMARY:
This study involves the use of an investigational drug called Creatine Monohydrate. This means that the drug has not yet been approved by the Food & Drug Administration (FDA) for treatment of altitude-induced depression. However, the FDA has not objected to its use to study its safety and effectiveness for preventing altitude-induced depression. This study will help find out what effects, good and/or bad, Creatine Monohydrate has on treating symptoms for altitude-induced depression. Creatine Monohydrate is believed to have an effect on improving symptoms of depression. The safety of Creatine Monohydrate in humans has been tested in prior research studies; however, some side effects may not yet be known.

DETAILED DESCRIPTION:
Subjects will be in this research study if they moved to Creech AFB from an elevation of less than 2.000 feet within the last month. The purpose of this study is to see if creatine monohydrate is effective in preventing altitude-induced depression. This study will enroll approximately 75 subjects.

This study involves the use of an investigational drug called Creatine Monohydrate. This means that the drug has not yet been approved by the Food & Drug Administration (FDA) for treatment of altitude-induced depression. However, the FDA has not objected to its use to study its safety and effectiveness for preventing altitude-induced depression. This study will help find out what effects, good and/or bad, Creatine Monohydrate has on treating symptoms for altitude-induced depression. Creatine Monohydrate is believed to have an effect on improving symptoms of depression. The safety of Creatine Monohydrate in humans has been tested in prior research studies; however, some side effects may not yet be known.

Creatine Monohydrate is a dietary supplement that is believed to aid in the building of muscle mass.

The placebo being used in this study is Maltodextrin (a sugar). Maltodextrin is an FDA approved food additive made from a highly processed starch product typically made from corn.

ELIGIBILITY:
PATIENTS MUST BE ABLE TO GET CARE AT NELLIS AIR FORCE BASE (A MILITARY INSTALLATION) IN ORDER TO PARTICIPATE IN THIS STUDY

Inclusion Criteria:

* Male and Female Active Duty members and DoD beneficiaries ages 18-65
* Moved to CREECH AFB from an altitude of less than 2,000 feet within the last month

Exclusion Criteria:

* Preexisting depression as noted in a review of their medical record or on their PHQ9 (score of 10 or greater)
* Preexisting anxiety as noted in a review of their medical record or on their GAD 7 (score of 10 or greater)
* Clinical or laboratory evidence of liver disease.
* Serum creatinine >1.5
* Existing kidney disease
* Existing Type I or Type II Diabetes Mellitus
* Taking creatine as a dietary supplement
* Moved to CREECH AFB from an altitude of greater than 2000 feet
* Pregnant, breast feeding, or trying to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 5 repeated measurements over the 120-day course of the study
  Questionnaire
Generalized Anxiety Disorder 7 (GAD-7) | 5 repeated measurements over the 120-day course of the study
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lee Church, MD, Principal Investigator — Mike O'Callaghan Military Medical Center
Locations (1):
- Mike O'Callaghan Military Medical Center, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):617-27. doi: 10.1001/archpsyc.62.6.617. PMID 15939839
- [Background] DelMastro K, Hellem T, Kim N, Kondo D, Sung YH, Renshaw PF. Incidence of major depressive episode correlates with elevation of substate region of residence. J Affect Disord. 2011 Mar;129(1-3):376-9. doi: 10.1016/j.jad.2010.10.001. Epub 2010 Nov 11. PMID 21074272
- [Background] Bardwell WA, Ensign WY, Mills PJ. Negative mood endures after completion of high-altitude military training. Ann Behav Med. 2005 Feb;29(1):64-9. doi: 10.1207/s15324796abm2901_9. PMID 15677302
- [Background] Lyoo IK, Yoon S, Kim TS, Hwang J, Kim JE, Won W, Bae S, Renshaw PF. A randomized, double-blind placebo-controlled trial of oral creatine monohydrate augmentation for enhanced response to a selective serotonin reuptake inhibitor in women with major depressive disorder. Am J Psychiatry. 2012 Sep;169(9):937-945. doi: 10.1176/appi.ajp.2012.12010009. PMID 22864465
- [Background] Armed Forces Health Surveillance Center (AFHSC). Absolute and relative morbidity burdens attributable to various illnesses and injuries, non-service member beneficiaries of the Military Health System, 2014. MSMR. 2015 Apr;22(4):27-34. No abstract available. PMID 25923401
- [Background] Brenner B, Cheng D, Clark S, Camargo CA Jr. Positive association between altitude and suicide in 2584 U.S. counties. High Alt Med Biol. 2011 Spring;12(1):31-5. doi: 10.1089/ham.2010.1058. Epub 2011 Jan 7. PMID 21214344
- [Background] Kim N, Mickelson JB, Brenner BE, Haws CA, Yurgelun-Todd DA, Renshaw PF. Altitude, gun ownership, rural areas, and suicide. Am J Psychiatry. 2011 Jan;168(1):49-54. doi: 10.1176/appi.ajp.2010.10020289. Epub 2010 Sep 15. PMID 20843869
- [Background] Drevets WC. Prefrontal cortical-amygdalar metabolism in major depression. Ann N Y Acad Sci. 1999 Jun 29;877:614-37. doi: 10.1111/j.1749-6632.1999.tb09292.x. PMID 10415674
- [Background] Rango M, Castelli A, Scarlato G. Energetics of 3.5 s neural activation in humans: a 31P MR spectroscopy study. Magn Reson Med. 1997 Dec;38(6):878-83. doi: 10.1002/mrm.1910380605. PMID 9402187
- [Background] Shi XF, Carlson PJ, Kim TS, Sung YH, Hellem TL, Fiedler KK, Kim SE, Glaeser B, Wang K, Zuo CS, Jeong EK, Renshaw PF, Kondo DG. Effect of altitude on brain intracellular pH and inorganic phosphate levels. Psychiatry Res. 2014 Jun 30;222(3):149-56. doi: 10.1016/j.pscychresns.2014.04.002. Epub 2014 Apr 13. PMID 24768210
- [Background] Lyoo IK, Kong SW, Sung SM, Hirashima F, Parow A, Hennen J, Cohen BM, Renshaw PF. Multinuclear magnetic resonance spectroscopy of high-energy phosphate metabolites in human brain following oral supplementation of creatine-monohydrate. Psychiatry Res. 2003 Jun 30;123(2):87-100. doi: 10.1016/s0925-4927(03)00046-5. PMID 12850248
- [Background] Poortmans JR, Francaux M. Adverse effects of creatine supplementation: fact or fiction? Sports Med. 2000 Sep;30(3):155-70. doi: 10.2165/00007256-200030030-00002. PMID 10999421
- [Background] Bizzarini E, De Angelis L. Is the use of oral creatine supplementation safe? J Sports Med Phys Fitness. 2004 Dec;44(4):411-6. PMID 15758854
- [Background] Edmunds JW, Jayapalan S, DiMarco NM, Saboorian MH, Aukema HM. Creatine supplementation increases renal disease progression in Han:SPRD-cy rats. Am J Kidney Dis. 2001 Jan;37(1):73-78. doi: 10.1053/ajkd.2001.20590. PMID 11136170
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Gadermann AM, Engel CC, Naifeh JA, Nock MK, Petukhova M, Santiago PN, Wu B, Zaslavsky AM, Kessler RC. Prevalence of DSM-IV major depression among U.S. military personnel: meta-analysis and simulation. Mil Med. 2012 Aug;177(8 Suppl):47-59. doi: 10.7205/milmed-d-12-00103. PMID 22953441